CLINICAL TRIAL: NCT03652142
Title: Predictive Biomarkers For Response To Nivolumab In Head and Neck Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, AMANDA PSYRRI, Medical Oncologist, Associate Professor, National Kapodistrian University of Athens, Attikon Hospital
Other Study IDs: CA209-8EN
Record Dates: First submitted 2018-06-20; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: HNSCC; DNA Damage; DNA Double Strand Break
Keywords: HNSCC; DDR; DNA damage; DNA damage repair; PD-L1; PD-1; NIVOLUMAB; Head and Neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Longitudinal tissue biopsies will be collected from HNSCC patients treated with nivolumab Biopsies will be taken at baseline, 24-72 hours after the second cycle of nivolumab and at progression.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Recurrent/metastatic HNSCC: The investigators will include recurrent/metastatic HNSCC patients who progressed after cisplatin-based chemotherapy and are to be treated with nivolumab. Tumor biopsies will be performed at baseline, after the second cycle and at progression with appropriate written informed consent and the samples will be analyzed. Biomarker research will be performed.
  The patients will receive intravenously nivolumab at dose of 240 mg every 2 weeks (240mg q2w). The patients will undergo tumor biopsy at baseline and within 24-72h after the second administration of treatment, and at progression of their disease.
  Interventions: Other: Biomarker Research; Drug: Nivolumab

INTERVENTIONS:
Other: Biomarker Research — The investigators will include recurrent/metastatic HNSCC patients who progressed after cisplatin-based chemotherapy and are to be treated with nivolumab 240mg IV q 2 weeks. Patient samples will be collected with appropriate written informed consent and analyzed.
Drug: Nivolumab — The investigators will include recurrent/metastatic HNSCC patients who progressed after cisplatin-based chemotherapy and are to be treated with nivolumab 240mg IV q 2 weeks.
  Other Names: Opdivo

SUMMARY:
Nivolumab is FDA-approved for the treatment of patients with recurrent/metastatic Head and Neck Squamous Cell Carcinoma (HNSCC).

HNSCC whose disease has progressed within 6 months after platinum-based chemotherapy. The development of predictive biomarkers is needed to optimize patient benefit, minimize risk of toxicities and guide combination strategies.

DETAILED DESCRIPTION:
Nivolumab is FDA-approved for the treatment of patients with recurrent/metastatic Head and Neck Squamous Carcinoma (HNSCC) whose disease has progressed within 6 months after platinum-based chemotherapy. The development of predictive biomarkers is needed to optimize patient benefit, minimize risk of toxicities and guide combination strategies. The greatest focus has been on tumor-cell programmed death Ligand 1 (PD-L1) expression. Although PD-L1 positivity enriches for populations with clinical benefit, PD-L1 testing alone is insufficient for patient selection in most malignancies. PD-L1 expression can be transient, and intrapatient and even intratumor heterogeneity in PD- L1 tumor expression can exist. Therefore, tumor sampling at one timepoint might not accurately reflect the state of PD1 axis in a patient. Another important aspect is that PD-L1 immunohistochemistry alone does not take into account factors that could impede the anti-PD1 therapy response such as whether or not active immune cell engagement of the PD1 axis occurs in the tumor microenvironment or other concurrent immune suppressive pathways are present.

Assessment of biomarkers at baseline may not predict benefit from immunotherapy. In a phase II study of ipilimumab in patients with metastatic melanoma baseline tumor infiltrating lymphocyte status was not associated with clinical activity. However, increase in tumor infiltrating lymphocyte density in tumor biopsy samples collected after the second dose of ipilimumab was associated with significantly greater clinical activity with ipilimumab compared to samples without increase in lymphocyte density. For a better understanding of the mechanisms of resistance to nivolumab in HNSCC, the investigators propose to study a cohort of longitudinal HNSCC samples from recurrent/metastatic HNSCC patients treated with nivolumab and identify biomarkers of response and resistance. The investigators will specifically focus on modulation of immune phenotype (ImmR) following two cycles of nivolumab as surrogate biomarker for response to nivolumab.

The primary endpoint will be the change in the percentage of immune cells that is caused by nivolumab treatment. Secondary endpoint will be safety of performing a biopsy after second nivolumab dose. Translational correlates will be tested in tumour tissue, plasma and germline DNA.

Investigator assessment of best overall response (BOR), determined between the date of first dose and the last tumor assessment (TA), will be image-based and scored using the RECIST 1.1. criteria. BOR will be defined as categorical variable with 3 levels { Benefit (complete response (CR), partial response (PR), stable disease (SD) lasting 6 months from the first nivolumab dose), no benefit (PD, progressive disease or SD lasting less than 6 months from the first nivolumab dose), and unknown} Longitudinal tissue biopsies will be collected from HNSCC patients treated with nivolumab . Biopsies will be taken at baseline, 24-72 hours after the second cycle of nivolumab and at progression.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any trial-related procedure is undertaken
* Male or female subjects aged ≥18 years
* Availability of a formalin-fixed, paraffin-embedded tissue sample (FFPE) containing tumor

Exclusion Criteria:

* no inform consent provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include recurrent/metastatic HNSCC patients who progressed after cisplatin-based chemotherapy and are to be treated with nivolumab.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of immune cells in post treatment compared to baseline biopsies | 2 weeks
  Primary endpoint will be the change in mean percentage of immune cells that is caused by the nivolumab treatment

SECONDARY OUTCOMES:
Safety of performing a biopsy after second nivolumab dose | 6 weeks
  Incidence of adverse events attributable to nivolumab treatment
Best overall response rate (BOR) according to RECIST 1.1 criteria | One year
  BOR will be defined as categorical variable with 3 levels { Benefit (complete response (CR), partial response (PR), stable disease (SD) lasting 6 months from the first nivolumab dose), no benefit (PD, progressive disease or SD lasting less than 6 months from the first nivolumab dose), and unknown}
Number of participants with tolerability to the treatment. | From the 1st day of therapy and every week for 4 weeks maximum and 30 days after last therapy administration ]
  NCI common toxicity criteria will be used
The burden of somatic non-synonymous mutations in association with BOR and survival | At baseline
  Targeted gene sequencing using next generation sequencing will be performed
The interferon-gamma gene signature in association with BOR and survival | At baseline
  Nanostring gene expression profiling, multiple tumor, inflammatory- and immune related genes will be analyzed by multiplex Nanostring technology by using the nCounter PanCancer Immune Profiling 770-plex gene expression Panel
The expression of PD-L1 in association with BOR and survival | At baseline and at 4 weeks
  PD-L1 will be assessed in tumor cells and immune cells by immunohistochemistry
The expression of human leukocyte antigens, HLA class I and HLA class II molecules in association with BOR and survival | At baseline
  It will be assessed at RNA and protein level
The presence of adaptive immunity cell populations | At baseline and at 4 weeks
  The assessment will be performed using multiplex imaging
The expression of PD-L2 in association with BOR and survival | At baseline and at 4 weeks
  PD-L2 will be assessed in tumor cells and immune cells by immunohistochemistry
PD-L1 expression in circulating tumor cells (CTCs) in association with BOR and survival | At baseline and at 4 weeks
  The assessment will be performed with Parsotrix system

CONTACTS AND LOCATIONS:
Overall Officials: AMANDA PSYRRI, MD, Principal Investigator — ATTIKON HOSPITAL, NATIONAL AND KAPODISTRIAN UNIVERSITY OF ATHENS, GREECE
Locations (1):
- Attikon Hospital, Athens, Chaidari, Greece

REFERENCES:
- [Background] Hamid O, Schmidt H, Nissan A, Ridolfi L, Aamdal S, Hansson J, Guida M, Hyams DM, Gomez H, Bastholt L, Chasalow SD, Berman D. A prospective phase II trial exploring the association between tumor microenvironment biomarkers and clinical activity of ipilimumab in advanced melanoma. J Transl Med. 2011 Nov 28;9:204. doi: 10.1186/1479-5876-9-204. PMID 22123319

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03652142/Prot_SAP_000.pdf